CLINICAL TRIAL: NCT06167330
Title: TITAN: a Randomised Controlled Trial Investigating the Effectiveness of Two Treatment Programs for Reducing Phantom Limb Pain Intensity and Its Interference with Function
Brief Title: TITAN Trial: Reducing Phantom Limb Pain in People with Amputations
Acronym: TITAN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Neuroscience Research Australia (Other)
Responsible Party: Principal Investigator, James McAuley, Principal Investigator, Neuroscience Research Australia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1296-2782; X23-0202 & 2023/ETH00540 (Other: RPAH Ethics and Governance Office)
Record Dates: First submitted 2023-11-26; First posted 2023-12-12 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Phantom Limb Pain; Amputation
MeSH Terms: conditions — Phantom Limb

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Progressive rehabilitation program (Experimental): The progressive rehabilitation program is a multicomponent intervention, including pain science education, sensory training, implicit and explicit motor imagery, and mirror therapy.
  Interventions: Other: Progressive rehabilitation program
- Stimulation devices (Experimental): The treatment program includes Transcutaneous Electrical Nerve Stimulation and Cranial Electrical Stimulation. Participants will complete activities at a self-directed pace following a standard progression protocol.
  Interventions: Other: Stimulation devices

INTERVENTIONS:
Other: Progressive rehabilitation program — Twelve-week treatment program delivered via eight, up to 1-hour telehealth sessions. The first five sessions will be scheduled every week, and the final three sessions will be scheduled fortnightly. Participants will also be prescribed approximately 15-30 minutes of home activities daily. The treatment program includes pain science education, sensory training, implicit and explicit motor imagery, and mirror therapy. Participants will complete activities at a self-directed pace following a standard progression protocol. Participant adherence will be measured via session attendance and self-report therapy diaries.
  Arms: Progressive rehabilitation program
Other: Stimulation devices — Twelve-week treatment program delivered via eight, up to 1-hour telehealth sessions. The first five sessions will be scheduled every week, and the final three sessions will be scheduled fortnightly. Participants will also be prescribed approximately 15-30 minutes of home activities daily. The treatment program includes transcutaneous electrical nerve stimulation and cranial electrical stimulation. Participants will complete activities at a self-directed pace following a standard progression protocol. Participant adherence will be measured via session attendance and self-report therapy diaries.
  Arms: Stimulation devices

SUMMARY:
The goal of this clinical trial is to investigate the effectiveness of two rehabilitation programs for individuals who have undergone amputations and are experiencing phantom limb pain. The main question it aims to answer is:

- In individuals who have undergone amputations and are experiencing phantom limb pain, what is the effectiveness of a progressive rehabilitation program compared to a treatment program consisting of transcutaneous electrical nerve stimulation and cranial electrical stimulation on reducing pain intensity and pain interference?

A total of 208 participants will be randomized into two groups: progressive rehabilitation program and stimulation devices. The progressive rehabilitation program includes pain science education, sensory training, and left/right judgements, imagined movements and mirror therapy. The treatment program for the group receiving the stimulation devices includes transcutaneous electrical nerve stimulation and cranial electrical stimulation. Both interventions will be delivered via eight, up to 1-hour telehealth sessions. Outcome measures will be assessed at baseline and weeks 12, 24 and 52.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing phantom limb pain for at least three months.
* Report at least one episode of phantom limb pain in the previous week.
* Report at least 4 points in pain intensity over the previous 7 days, assessed using the 11-point Numerical Pain Rating Scale.
* Be a resident in Australia for the intervention and follow-up period.
* Have access to the internet and smart device (e.g., mobile phone).
* Be proficient in English.

Exclusion Criteria:

* Bilateral amputation.
* Scheduled for major surgery during the study period.
* Pain in the intact limb.
* Vision impairment that would preclude successful participation.
* Auditory impairment that would preclude successful participation.
* Cognitive problems that would preclude effective participation in trial procedures (e.g., Alzheimer's, dementia).
* Previously diagnosed neurological disorders that affect the movement of the intact limb (e.g., stroke, Parkinson, Multiple Sclerosis).
* Completed Graded Motor Imagery in the order of left/right judgements, imagined movements, and mirror therapy.
* Have contraindications for the use of stimulation devices (e.g., pacemaker, spinal cord stimulator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-12-18 (Estimated); Study Completion 2027-12-18 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Week 12 post-randomisation
  Average pain intensity over the previous 7 days assessed using the 11-point Numerical Pain Rating Scale.
Pain interference | Week 12 post-randomisation
  Average pain interference with function over the previous 7 days assessed using the 0-10 Pain Interference Scale of the Brief Pain Inventory.

SECONDARY OUTCOMES:
Pain intensity | Weeks 24 and 52 post-randomisation
  Average pain intensity over the previous 7 days assessed using the 11-point Numerical Pain Rating Scale.
Pain interference | Weeks 24 and 52 post-randomisation
  Average pain interference with function over the previous 7 days assessed using the 0-10 Pain Interference Scale of the Brief Pain Inventory.
Pain severity | Weeks 12, 24 and 52 post-randomisation
  Average pain intensity over the previous 7 days assessed using the 0-10 Pain Severity Scale of the Brief Pain Inventory.
Sleep subscale of the Brief Pain Inventory's Pain Interference Scale | Weeks 12, 24 and 52 post-randomisation
  Sleep Quality assessed using the Sleep subscale of the Brief Pain Inventory's Pain Interference Scale. The participants will rate the interference of pain with sleep on a 0-10 scale where "0" represents "does not interfere" and "10" represents "completely interferes".
PROMIS Self-Efficacy Manage Symptoms | Weeks 12, 24 and 52 post-randomisation
  Pain Self-efficacy assessed using PROMIS Self-Efficacy Manage Symptoms (Computer Adaptive Test) (28-item version; higher scores mean more self-efficacy).
PROMIS Depression | Weeks 12, 24 and 52 post-randomisation
  Emotional distress and depression assessed using PROMIS Depression (Computer Adaptive Test) (28-item version; higher scores mean more depression).
EuroQol 5-Dimension 5-Level (EQ-5D-5L) | Weeks 12, 24 and 52 post-randomisation
  Health-Related Quality of Life assessed using the EQ-5D-5L dimensions scale range, 1-5; higher scores indicate better quality of life) and health thermometer (range, 0-100; higher scores indicate better quality of life).
Global Perceived Effect Scale | Weeks 12, 24 and 52 post-randomisation
  Perception of recovery assessed using the Global Perceived Effect scale (range from -5 to +5; higher scores mean greater improvement).
Adverse events | From randomisation to week 12 post-randomisation
  Adverse events assessed via self-report.
Adherence to treatment | From randomisation to week 12 post-randomisation
  Adherence to treatment assessed via session attendance and self-report (diary), including frequency per week and duration per day.
Total health-care costs | Weeks 12, 24 and 52 post-randomisation
  Total health-care costs will be estimated as the trial intervention costs and outside trial health-care resource use attributable to phantom limb pain from the Medicare Benefits Scheme and Pharmaceutical Benefits Scheme. Quality-adjusted life-years (QALYs) from the EQ-5D-5L using the Australian utility weights will also be used in the trial-based cost-utility analysis.
Treatment rationale credibility | Week 1 post-randomisation
  Treatment rationale credibility assessed using the Credibility and Expectancy Questionnaire. The total score ranges from 0 to 48, with lower scores indicating lower credibility.

OTHER OUTCOMES:
Pain Self-Efficacy Questionnaire (mediator) | Weeks 6 and 10 post-randomisation
  Pain self efficacy measured using the Pain Self-Efficacy Questionnaire. The total score of this questionnaire ranges from 0 to 60, with higher scores indicating higher self-efficacy and functioning despite ongoing pain.
Concept of Pain Inventory (mediator) | Weeks 6 and 10 post-randomisation
  Beliefs and knowledge of pain science assessed using the Concept of Pain Inventory. This is a 13-item questionnaire with scores ranging from 0 to 52 points, with higher scores reflecting greater alignment with contemporary pain science.
Pain Catastrophising Scale (mediator) | Weeks 6 and 10 post-randomisation
  Pain catastrophising assessed using the Pain Catastrophising Scale. The total score ranges from 0 to 52, with higher scores indicating a higher level of catastrophising.
Phantom limb movement scale (mediator) | Weeks 6 and 10 post-randomisation
  The ability to move the phantom limb assessed on an 11-point Numerical Rating Scale (0: No movement at all, 10: Complete range of movement as if the limb were still present).
Phantom limb body perception disturbance scale (mediator) | Weeks 6 and 10 post-randomisation
  The phantom limb body perception disturbances assessed using 4 questions measuring ownership, awareness, attention and emotional feelings on an 11-point Numerical Rating Scale (range, 0-40; lower scores indicate more severe body perception disturbances). Adapted from the Bath Complex Regional Pain Syndrome body perception disturbance scale.

CONTACTS AND LOCATIONS:
Overall Officials: James H McAuley, PhD, Principal Investigator — Neuroscience Research Australia
Locations (1):
- Neuroscience Research Australia, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be made to interested researchers only upon reasonable request and once the proposed research project has received separate ethics approval from a Human Research Ethics Committee.
  Request to the data custodian, the Principal Investigator (j.mcauley@neura.edu.au).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available after the publication of study reports. There is no end date for the availability of study data.

REFERENCES:
- [Background] Limakatso K, Cashin AG, Williams S, Devonshire J, Parker R, McAuley JH. The Efficacy of Graded Motor Imagery and Its Components on Phantom Limb Pain and Disability: A Systematic Review and Meta-Analysis. Can J Pain. 2023 May 17;7(1):2188899. doi: 10.1080/24740527.2023.2188899. eCollection 2023. PMID 37214633
- See also: Trial website — https://titan.neura.edu.au/